CLINICAL TRIAL: NCT01754701
Title: Acute vs. Delayed Iron: Effect on Red Cell Iron Incorporation in Severe Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1203M11234; 1R03HD074262 (NIH)
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Iron Deficiency; Malaria; Nutrition; Global Health
MeSH Terms: conditions — Iron Deficiencies; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate iron (Experimental): Children who start 4 weeks of iron therapy on Day 0
  Interventions: Dietary Supplement: Immediate iron
- Delayed iron (Experimental): Children who start 4 weeks of iron therapy on Day 28
  Interventions: Dietary Supplement: Delayed iron

INTERVENTIONS:
Dietary Supplement: Immediate iron — Children who start 4 weeks of iron therapy on Day 0
  Other Names: Ferrous sulfate syrup
  Arms: Immediate iron
Dietary Supplement: Delayed iron — Children who start 4 weeks of iron therapy on Day 28
  Arms: Delayed iron

SUMMARY:
The purpose of this study is to determine whether iron therapy given to iron-deficient Ugandan children with moderate-to-severe anemia and clinical malaria is better absorbed and incorporated into red blood cells if it is given concurrently with antimalarial treatment on Day 0 (immediate group) or 4 weeks after antimalarial treatment on Day 28 (delayed group). Use of iron stable isotopes 57Fe and 58Fe will permit measurement of red blood cell iron incorporation on Day 0 and Day 28 in all children. The investigators hypothesize that red cell iron incorporation at the time of initial supplement administration will be greater in children receiving delayed vs. immediate iron (Aim 1), and children in the delayed group will also have greater hematological recovery on Day 56 than children in the immediate group (Aim 2).

DETAILED DESCRIPTION:
Approximately 1 million children < 5 y living in sub-Saharan Africa die from severe anemia annually. This severe anemia frequently results from coexisting iron deficiency and malaria infection, but the standard of care, concurrent iron therapy and antimalarial treatment, has proven ineffective at curing the profound anemia and has promoted proliferation of the parasite in some studies. The pro-inflammatory immune response mounted against malaria down-regulates iron absorption in the gut, making provision of oral iron supplements during malarial infection of questionable utility. The present study proposes to use iron stable isotopes and a randomized design to test whether starting 4 weeks of iron therapy immediately after antimalarial treatment or 4 weeks later is associated with greater iron incorporation into red blood cells at the time of initial administration of iron therapy and improved long-term hematological recovery. One hundred severely anemic (hemoglobin 5-9.9 g/dL) Ugandan children 6-59 mos with clinical signs of malaria who present to the Pediatric Acute Care Ward of Mulago Hospital in Kampala, Uganda, will be randomized to start iron immediately after antimalarial treatment on Day 0 (immediate group) or 4 weeks later on Day 28 (delayed group). Children will be assessed at the hospital on Day 0, Day 28 and Day 56 and will receive bi-weekly home visits for the 56-day study duration. The specific aims and corresponding hypotheses of the proposed study are:

Aim 1: Identify the sequencing of antimalarial treatment and iron therapy that results in the greatest red cell iron incorporation at the time of initial iron supplement administration. The working hypothesis is that red cell iron incorporation will be greater at the time of initial supplement administration in children starting iron 4 weeks after antimalarial treatment (delayed group) compared to children starting iron concurrently with antimalarial treatment (immediate group), due to more complete parasite clearance and resolution of inflammation, permitting better iron uptake, distribution, and utilization.

Aim 2: Determine whether long-term hematological recovery is impacted by immediate vs. delayed iron. The working hypothesis is that delayed iron treatment will be associated with greater hemoglobin and improved iron status at Day 56 compared to immediate treatment due to more complete parasite clearance and consequent improved iron absorption and use in the delayed group.

The results of this study will establish a physiologically-based framework for the optimal timing of antimalarial treatment and iron therapy upon which future interventions aimed at improving iron status in malaria-endemic regions can be built, thus helping to reduce the morbidity and mortality and ensure the full neurobehavioral development of the millions of severely anemic children suffering from iron-deficiency and malaria.

ELIGIBILITY:
Inclusion Criteria:

1. 6 - 59 months of age
2. Hemoglobin 5.0 - 9.9 g/dL according to HemoCue
3. Temperature > 37.5°C or history of fever in past 24 hours
4. P. falciparum on blood smear at Acute Care Unit
5. Residence<50 km of study hospital

Exclusion Criteria:

1. Impaired consciousness on physical exam or history of coma with present illness
2. Seizure activity prior to or during admission
3. Known sickle cell disease 4) Acute malnutrition

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percent red blood cell iron incorporation on Day 0 in children in the immediate group vs. percent red blood cell iron incorporation on Day 28 in children in the delayed group | 56 days
  All children will receive iron stable isotope 57Fe on Day 0 and iron stable isotope 58Fe on Day 28. Children in the immediate group will begin 27 days of daily iron syrup at home on Day 1. Children in the delayed group will begin 27 days of daily iron syrup at home on Day 29. All children will be assessed at the hospital at Day 28 and Day 56.

SECONDARY OUTCOMES:
Hematological recovery in the immediate vs. delayed groups on Day 56 | 56 days
  All children will receive iron stable isotope 57Fe on Day 0 and iron stable isotope 58Fe on Day 28. Children in the immediate group will begin 27 days of daily iron syrup at home on Day 1. Children in the delayed group will begin 27 days of daily iron syrup at home on Day 29. All children will be assessed at the hospital at Day 28 and Day 56.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cusick, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Cusick SE, Opoka RO, Abrams SA, John CC, Georgieff MK, Mupere E. Delaying Iron Therapy until 28 Days after Antimalarial Treatment Is Associated with Greater Iron Incorporation and Equivalent Hematologic Recovery after 56 Days in Children: A Randomized Controlled Trial. J Nutr. 2016 Sep;146(9):1769-74. doi: 10.3945/jn.116.233239. Epub 2016 Jun 29. PMID 27358418